CLINICAL TRIAL: NCT04104802
Title: Study of the Facial Nerve in MRI 3T in the Preoperative Assessment of Parotid Tumors
Acronym: FACPAR
Status: Withdrawn | Type: Observational
Why Stopped: refusal of the ansm
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ACN_2019_12
Record Dates: First submitted 2019-06-24; First posted 2019-09-26 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Parotid Tumor
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — All patients included will benefit from both methods of assessing anatomical relationships between the facial nerve and the parotid tumor:
  1) New medical imaging technique evaluated: 3 Tesla Parotidic MRI High Resolution with Specific Sequences and Gadolinium Injection 2) Standard Gold: Intraoperative Exam

SUMMARY:
Preoperative evaluation of the precise localization of the intrapartotic facial nerve is essential for the ENT surgeon to assess the risk of nerve damage during parotid tumor excision, and inform the patient of the risk of post-paralyzed facial nerve palsy. procedure

DETAILED DESCRIPTION:
1. st visit: Inclusion, parotid MRI 3Tesla high resolution with specific sequences and gadolinium injection performed at the A. de Rothschild Foundation. Evaluation by two radiologists of the exact position of the parotid tumor with respect to the trunk of the facial nerve and its first branches, classified into two categories: contact (≤ 5 mm) or distance (> 5 mm).
2. nd visit: Surgical intervention of the parotid tumor. The surgeon will specify the same data as those collected by the radiologists after the MRI. The surgeon will not be aware of the data concerning the ratios of parotid tumor to facial nerve collected on MRI sequences for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient seeking first-line surgery for a parotid tumor (single or multiple, benign or malignant)
* Parotidian tumor located near the trunk of the facial nerve and / or its first division branches (temporofacial and cervicofacial), during a clinical evaluation performed by the surgeon in preoperative consultation
* Patient affiliated or beneficiary of a social security scheme
* Written consent to participate in the study

Exclusion Criteria:

* Personal history of ipsilateral parotid surgery
* Contraindication to MRI (electronic device, metallic foreign body, claustrophobia)
* Known hypersensitivity to gadolinium contrast agents
* Renal impairment known: glomerular filtration rate <30 mL / min
* Pre or post-operative period of liver transplantation
* Patient benefiting from a legal protection measure
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient candidate for first-line surgery for a parotid tumor
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity of a high-resolution 3 Tesla MRI with gadolinium injection with specific sequences versus intraoperative findings of the surgeon (gold standard), to evaluate the anatomic relationships between parotid tumor and facial nerve. | 1 day
  Sensitivity of new MRI sequences to determine whether the parotid tumor is in contact or at a distance from the facial nerve (common core and first division branches) in comparison with the intra-operative examination (gold standard).
  The contact between the parotid tumor and the trunk of the facial nerve or its first branches of division is a binary qualitative variable with modalities defined as:
  * "Yes": tumor on contact (distance between the tumor and the trunk of the facial nerve or its first branches between 0 and 5 mm)
  * "No": trunk of the facial nerve or its first divisional branches located at a distance (ie more than 5mm from the parotid tumor).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Fondation Adolphe De Rothschild, Paris
  - Hôpital Saint Joseph, Paris
  - Institut Arthur Vernes, Paris
  - Hôpital FOCH, Suresnes